CLINICAL TRIAL: NCT01167400
Title: Cybercycling for Older Adults: Neuropsychological, Physiological and Behavioral Effects
Brief Title: Cybercycling for Cognitive Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Union College, New York (Other)
Collaborators: Skidmore College (Other)
Responsible Party: Principal Investigator, Cay Anderson-Hanley, Associate Professor, Union College, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS1259; 64449 (Other Grant/Funding Number: Robert Wood Johnson Foundation)
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Cognitive Ability, General
Keywords: exercise; executive function; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cybercycling (Experimental): cybercycling for 3 months
  Interventions: Behavioral: Cybercycling
- Traditional Stationary Biking (Active Comparator): Traditional exercise on a stationary bike for 3 months.
  Interventions: Behavioral: Traditional exercise

INTERVENTIONS:
Behavioral: Cybercycling — exercising on a videogame-enhanced interactive 3D stationary bicycle for 3 months, 3-5x/wk
  Other Names: Netathalon; Expresso
  Arms: Cybercycling
Behavioral: Traditional exercise — exercising on a traditional stationary bike for 3 months, 3-5x/wk
  Other Names: Tunturi
  Arms: Traditional Stationary Biking

SUMMARY:
Exercise has been linked to cognitive health, but few older adults exercise at recommended levels. Cybercycling may provide additional cognitive benefits due to increased motivation to ride the interactive 3D tours. Participants will be randomly assigned to three months of either cybercycling or traditional stationary biking; and they will complete comprehensive evaluations before and after exercise. Older adults are expected to show significant neuropsychological, physiological and behavioral gains.

DETAILED DESCRIPTION:
The purpose of this study is to test the following hypotheses: (1) stationary cycling with virtual reality tours ("cybercyle") will enhance executive function and clinical status more than traditional exercise; (2) exercise effort will explain improvement; and (3) brain-derived neurotrophic growth factor (BDNF) will increase.

ELIGIBILITY:
Inclusion Criteria:

* age 50+
* able to participate in cycling
* physician permission

Exclusion Criteria:

* unstable heart condition
* physician denial
* neurological condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function after three months of exercise. | 3 months
  Cognitive function, especially executive function, will be assessed before and after three months of either cybercycling or traditional exercise biking. Neuropsychological tests will assess: cognitive flexibility and simultaneous processing(i.e., Stroop, Digits Backwards, and Trails Difference Score).

SECONDARY OUTCOMES:
Weight | 3 months
  Weight and other physiological factors will be assessed before and after 3 months of exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — Union College; Paul Arciero, DPE, Principal Investigator — Skidmore College
Locations (8):
- United States (8):
  - Beltrone Living Center, Colonie, New York
  - Highpointe Apartments, Malta, New York
  - Glen Eddy, Niskayuna, New York
  - Prestwick Chase, Saratoga Springs, New York
  - Wesley Health Care (Woodlawn and Embury), Saratoga Springs, New York
  - Westview Apartments, Saratoga Springs, New York
  - Kingsway Village, Schenectady, New York
  - Schaffer Heights, Schenectady, New York

REFERENCES:
- [Result] Anderson-Hanley C, Arciero PJ, Brickman AM, Nimon JP, Okuma N, Westen SC, Merz ME, Pence BD, Woods JA, Kramer AF, Zimmerman EA. Exergaming and older adult cognition: a cluster randomized clinical trial. Am J Prev Med. 2012 Feb;42(2):109-19. doi: 10.1016/j.amepre.2011.10.016. PMID 22261206